CLINICAL TRIAL: NCT02030574
Title: BrUOG 300: Neoadjuvant Gemcitabine and Fractionated, Weekly Cisplatin For Muscle Invasive Bladder Cancer and Patients Not Candidates For High Dose Cisplatin
Brief Title: Neoadjuvant Gemcitabine and Fractionated, Weekly Cisplatin For Muscle Invasive Bladder Cancer and Patients Not Candidates For High Dose Cisplatin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study is being closed to accrual secondary to low accrual and an interest in opening up a different trial.
Sponsor: Brown University (Other)
Collaborators: Lifespan (Other)
Responsible Party: Principal Investigator, Jodi Layton, Principal Investigator, Brown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 300
Record Dates: First submitted 2013-12-20; First posted 2014-01-08 (Estimated); Results first posted 2016-03-25 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-07

CONDITIONS: Invasive Bladder Cancer; Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine and fractionated cisplatin (combination treatment) (Experimental): 1 Cycle = 21 days. GC x 4 cycles ----> cystectomy Gemcitabine: 1000mg/m2, days 1 and 8 Cisplatin: 35mg/m2, days 1 and 8
  Interventions: Drug: Gemcitabine and fractionated cisplatin (combination treatment)

INTERVENTIONS:
Drug: Gemcitabine and fractionated cisplatin (combination treatment) — 1 Cycle = 21 days. GC x 4 cycles ----> cystectomy Gemcitabine: 1000mg/m2, days 1 and 8 Cisplatin: 35mg/m2, days 1 and 8

SUMMARY:
The standard treatment of muscle invasive bladder cancer is to administer chemotherapy for approximately 3 months then to have surgery to remove the bladder. Chemotherapy may reduce the size of the cancer in your bladder before surgery and can also help to reduce the chance that your bladder cancer will come back (metastasize) in other parts of your body after bladder surgery.

This study will involve testing cisplatin in lower weekly doses with gemcitabine.The purpose of this study is to test the effects, good and bad, of low dose weekly cisplatin and gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed muscle-invasive urothelial (transitional cell) carcinoma of the bladder or upper genitourinary tract.
2. Stage T2-T4a. Patients may have nodal disease but there must be no evidence of distant metastases and patients must be candidates for radical cystectomy as determined by urologic surgeon (note from/confirmation by surgeon required).
3. No prior systemic therapy for urothelial carcinoma. Prior intravesical therapy is allowed.
4. Patients are determined by their treating oncologist to not be a candidate high dose cisplatin (> 70mg/m2) due to medical comorbidities.
5. Creatinine Clearance (CrCL or eCCr)) > 25 mL/min calculated using the Cockcroft-Gault formula
6. Patients without serious medical risk factors involving any of the major organ systems such that the investigator considers it unsafe for the patient to receive the protocol treatment of this study with gemcitabine and weekly fractionated cisplatin.
7. Preexisting neuropathy < grade 2.
8. No prior invasive malignancy within the prior two years. However, prior history of non-muscle invasive bladder cancer and patients with an early stage malignancy that is not expected to require treatment in the next 2 years (such as early stage, resected breast cancer, or asymptomatic prostate cancer) are eligible.
9. ECOG performance status 0 or 1.
10. Age ≥ 18 years of age.
11. Not pregnant and not nursing. Women of child bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to beginning of treatment. Post-menopausal women (surgical menopause or lack of menses >12 months) do not need to have a pregnancy test, please document status.
12. Required Initial Laboratory Values:

    * Neutrophils ≥ 1,000/μl
    * Platelet count ≥ 100,000/μl
    * Total bilirubin ≤ 1.5 x ULN.
    * AST (SGOT) & ALT (SGPT) ≤ 3.0 x ULN

Exclusion Criteria:

1. Metastatic disease.
2. Prior hypersensitivity to platinums that in the investigators opinion would put the patient at risk if re-exposed
3. Small cell cancer of the bladder or pure adenocarcinoma. Patients with mixed histologies such as urothelial carcinoma with sarcomatoid features, squamous differentiation or adenocarcinoma are allowed as long as transitional cell cancer is the predominant pathologic subtype.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rhode Island Hospital (including Newport Hospital and East Greenwich), Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine and Fractionated Cisplatin (Combination Treatment): 1 Cycle = 21 days. GC x 4 cycles ----> cystectomy Gemcitabine: 1000mg/m2, days 1 and 8 Cisplatin: 35mg/m2, days 1 and 8
  Gemcitabine and fractionated cisplatin (combination treatment): 1 Cycle = 21 days.
  GC x 4 cycles ----> cystectomy Gemcitabine: 1000mg/m2, days 1 and 8 Cisplatin: 35mg/m2, days 1 and 8
Period: Overall Study
Arm/Group | Gemcitabine and Fractionated Cisplatin (Combination Treatment)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine and Fractionated Cisplatin (Combination Treatment)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 63.5 [51 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate of Neoadjuvant Gemcitabine and Fractionated Cisplatin for Patients With Muscle Invasive Bladder Cancer Whom Are Not Candidates for High Dose Cisplatin.
Description: Response will be evaluated in this study using the international criteria proposed in the Revised Response Evaluation Criteria in Solid Tumors (RECIST) Guideline version 1.1 [Eur J Cancer. 2009;45:228-247.].Complete Response (CR): Disappearance of all target lesions; Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficie
Time Frame: at approximately 6 months
Measure: Number; unit: participants
Arm/Group | Gemcitabine and Fractionated Cisplatin (Combination Treatment)
Number analyzed (Participants) | 2
participants | 2

2. Secondary Outcome: Number of Participants Experiencing Toxicities With Neoadjuvant Gemcitabine and Fractionated Cisplatin for Patients With Bladder Cancer
Description: Toxicities assessed while patients are on treatments
Time Frame: Prior to each of the 4 cycles of treatment, after 4 months of treatment, 30 days post the last dose of drug (for a total of approximately 5 months)
Measure: Number; unit: participants
Arm/Group | Gemcitabine and Fractionated Cisplatin (Combination Treatment)
Number analyzed (Participants) | 2
participants | 2

ADVERSE EVENTS:
Time Frame: Prior to each of the 4 cycles of treatment, after 4 months of treatment, 30 days post the last dose of drug (for a total of approximately 5 months)
Arm/Group | Gemcitabine and Fractionated Cisplatin (Combination Treatment)
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine and Fractionated Cisplatin (Combination Treatment) (N=2)
thromboembolic event and pain right arm (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine and Fractionated Cisplatin (Combination Treatment) (N=2)
phlebitis (Blood and lymphatic system disorders) | 1 (1)
urinary frequency (Gastrointestinal disorders) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Platelet Count (Blood and lymphatic system disorders) | 2 (2)
Sodium (Blood and lymphatic system disorders) | 2 (2)
Hemaglobin/anemia (Blood and lymphatic system disorders) | 1 (1)
Absolute Neutrofil Count (Blood and lymphatic system disorders) | 1 (1)
epistaxis (Blood and lymphatic system disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
joint knee swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
facial flushing (Blood and lymphatic system disorders) | 1 (1)
Magnesium (Blood and lymphatic system disorders) | 1 (1)
pain (General disorders) | 1 (1)
urinary incontinence (Gastrointestinal disorders) | 1 (1)
abdomnial pain (General disorders) | 1 (1)
Acute Kidney Infection (Gastrointestinal disorders) | 1 (1)
hydronephrosis (urostomy obstruction) (Gastrointestinal disorders) | 1 (1)
lymphocele (Investigations) | 1 (1)
cough (General disorders) | 2 (2)
dyspnea/Shorness Of Breath (Cardiac disorders) | 1 (1)
Urinary Track Infection (Investigations) | 1 (1)
Sepsis (Blood and lymphatic system disorders) | 1 (1)
pulmonary embolism (Blood and lymphatic system disorders) | 1 (1)
Albumin (Blood and lymphatic system disorders) | 1 (1)
Potassium (Blood and lymphatic system disorders) | 1 (1)
persistent urine leak (moderate per site not a gradable event)(pt 1) (Gastrointestinal disorders) | 1 (1)
abd fluid collection (moderate per site not a gradable event)(pt 1) (General disorders) | 1 (1)
decreased urine drainage ( mild per site not a gradeable event)(pt 1) (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study has been terminated secondary to low accrual and an interest in opening up a different trial; more tailored to Physician interests and patient need.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No